CLINICAL TRIAL: NCT02364752
Title: A Clinical Trial to Evaluate Circulating and Imaging Biomarkers in Heart Failure Patients
Brief Title: A Study Evaluating Biomarkers in Participants With Heart Failure (MK-0000-344)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-344
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy (Experimental): Part 1: Blood is obtained from healthy participants on 3 consecutive days, and participants undergo Cardiac Magnetic Resonance Imaging (CMR) and two-dimensional speckle tracking echocardiography (2DSTE) on one of those 3 days.
  Interventions: Procedure: Blood Draw
- Mild/moderate heart failure (HF) (Experimental): Part 1: Blood is obtained from participants with mild/moderate HF on 3 consecutive days, and participants undergo CMR and 2DSTE on one of those 3 days. Part 2: Within 5 days of completing Part 1 participants have a 24 hour loop diuretic withdrawal, and 15 hour 0.9% normal saline infusion; followed by a blood draw, CMR and 2DSTE.
  Interventions: Procedure: Blood Draw; Procedure: Loop Diuretic Withdrawal/Salt Load
- Severe HF (Experimental): Part 1: Blood is obtained from participants with severe HF on 3 consecutive days, and participants undergo CMR and 2DSTE on one of those 3 days. Part 2: Within 5 days of completing Part 1 participants have a 24 hour loop diuretic withdrawal, and 15 hour 0.9% normal saline infusion; followed by a blood draw, CMR and 2DSTE.
  Interventions: Procedure: Blood Draw; Procedure: Loop Diuretic Withdrawal/Salt Load

INTERVENTIONS:
Procedure: Blood Draw
Procedure: Loop Diuretic Withdrawal/Salt Load
  Arms: Mild/moderate heart failure (HF); Severe HF

SUMMARY:
The aim of this 2-part study is to assess B-type natriuretic peptide (BNP) as well as other circulating and imaging biomarkers in myocardial function. Part 1 assesses biomarker levels in healthy participants and participants with cardiac dysfunction. Part 2 assesses BNP and other circulating biomarker levels, and performs imaging in participants with cardiac dysfunction who continued from Part 1. The primary hypothesis is that compared to healthy participants, biomarker levels are elevated in participants with mild/moderate and severe cardiac dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* female of reproductive potential must demonstrate non-pregnant state, and agree to use two acceptable methods of birth control
* postmenopausal or surgically sterile female
* have a Body Mass Index (BMI) >= 18 and =< 35 kg/m^2, inclusive
* healthy participants are in general good health
* participants with HF have no untreated, significant health issue from other co-morbidities, e.g. uncontrolled hypertension
* is willing to undergo echocardiography, CMR, and other study assessments
* participants with HF have a diagnosis of cardiomyopathy, and slight to moderate limitation of physical activity, but are comfortable at rest
* participants with HF are on a stable medical therapy for HF for two weeks prior to start of Part 1
* participants with HF are on a stable diuretic regimen of >= 40 mg/day furosemide or >= 10 mg/day torsemide for at least 2 weeks prior to start of Part 1

Exclusion Criteria:

* has any clinically significant, uncontrolled renal, endocrine (except Type II Diabetes), neurological, hepatic, immunological or inflammatory disease
* has a history of cancer (malignancy)
* had major surgery or donated/lost approximately 500 mL of blood within 4 weeks prior to screening
* participated in another investigational trial within 4 weeks prior to screening
* excepting permitted medications, uses prescription, or non-prescription drugs or herbal remedies 2 weeks prior to enrollment until completion of trial
* takes medications that affect BNP levels within 30 days prior to screening
* undergoes high-intensity physical exercise from 1 week prior to pretrial visit until completion of trial
* has implanted or embedded metal objects in body that in response to a magnetic field could cause injury
* suffers from claustrophobia making them unable to undergo CMR scanning
* consumes alcohol for 7 days prior to screening until completion of study
* consumes excessive amounts of caffeinated beverages
* uses cannabis regularly, or any illicit drugs, or has a history of drug (including alcohol) abuse within prior 12 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Level of total BNP in Part 1 | Up to Day 3
Level of total BNP in Part 2 | Up to Day 1 post-loop diuretic withdrawal (Up to Day 10)

SECONDARY OUTCOMES:
Level of active BNP in Part 1 | Up to Day 3
Level of active BNP in Part 2 | Up to Day 1 post-loop diuretic withdrawal (Up to Day 10)
Ratio of total BNP/active BNP in Part 1 | Up to Day 3
Ratio of total BNP/active BNP in Part 2 | Up to Day 1 post-loop diuretic withdrawal (Up to Day 10)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC